CLINICAL TRIAL: NCT03262766
Title: Daily Intermittent Hypoxia and Task-Specific Upper Limb Training in Persons With Chronic Incomplete SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STU00204305; 81428 (Other Grant/Funding Number: Midwest Regional Spinal Cord Injury Care System grant); 81349 (Other Grant/Funding Number: National Institute on Disability and Rehabilitation Research)
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
Keywords: Acute Intermittent Hypoxia; Upper Extremity Training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Subjects will then be randomized to one of the four arms. The four arms of interventions are:
  1. Acute intermittent hypoxia (AIH) therapy
  2. AIH therapy + Upper extremity training
  3. Sham AIH therapy + Upper extremity training
  4. Sham Hypoxia
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a blinded study, which means the participant will not know which treatment they are receiving. They will either receive intermittent periods of low oxygen (hypoxia) or a session composed of only normal room air. They will be randomly assigned to a treatment based on chance, like a flip of a coin. Neither you nor the researcher chooses your assigned group. They will have an equal chance of being in either group. Upon acceptance into the study, subjects will be assigned an identification number. Data pertaining to each subject will only be identified by this number. Any forms/files containing the subject's personal information and their ID number will be housed in a locked office/laboratory space. The outcomes assessor will also be blinded to the intervention the subject received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acute intermittent hypoxia (AIH) (Active Comparator): Subjects will be exposed to acute intermittent hypoxia, daily for 5 days. Each session will consist of up to 90 seconds of 9-10% Oxygen (FiO2 0.09), alternating with up to 90 seconds of 21% Oxygen (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for up to 45 minutes, to maintain SpO2 at 80-90%. If the SpO2 drops below 75%, hypoxia exposure will be terminated immediately.
  There is continuous monitoring of respiratory rate, heart rate and peripheral arterial oxyhemoglobin saturation (SpO2).
  Interventions: Other: Acute Intermittent Hypoxia (AIH)
- AIH+ Upper extremity training (Experimental): Subjects will be exposed to acute intermittent hypoxia, daily for 5 days. Each session will consist of up to 90 seconds of 9-10% Oxygen (FiO2 0.09), alternating with up to 90 seconds of 21% Oxygen (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for up to 45 minutes, to maintain SpO2 at 80-90%. If the SpO2 drops below 75%, hypoxia exposure will be terminated immediately.
  There is continuous monitoring of respiratory rate, heart rate and peripheral arterial oxyhemoglobin saturation (SpO2).
  Following the AIH protocol, subjects will receive 45 minutes of task-specific, high repetition upper extremity training, given using an upper-limb robotic rehabilitation device, the Armeo Spring®.
  Interventions: Other: Acute Intermittent Hypoxia (AIH); Behavioral: Upper extremity training
- Sham AIH + Upper extremity training (Active Comparator): Subjects will be exposed to sham hypoxia daily for 5 days. Each session will consist of up to 90 seconds of 21% Oxygen (FiO2 0.21), alternating with up to 90 seconds of 21% Oxygen (normoxic air FiO2 0.21). The delivery will be repeated up to 18 times per session each, for a total of up to 45 minutes.
  There is continuous monitoring of respiratory rate, heart rate and peripheral arterial oxyhemoglobin saturation (SpO2).
  Following the sham AIH protocol, subjects will receive 45 minutes of task-specific, high repetition upper extremity training. Upper extremity training will be given using an upper-limb robotic rehabilitation device, the Armeo Spring®.
  Interventions: Behavioral: Upper extremity training; Other: Sham Acute intermittent hypoxia
- Sham Acute intermittent hypoxia (Sham Comparator): Subjects will be exposed to sham hypoxia daily for 5 days. Each session will consist of up to 90 seconds of 21% Oxygen (FiO2 0.21), alternating with up to 90 seconds of 21% Oxygen (normoxic air FiO2 0.21). The delivery will be repeated up to 18 times per session each, for a total of up to 45 minutes.
  There is continuous monitoring of respiratory rate, heart rate and peripheral arterial oxyhemoglobin saturation (SpO2).
  Interventions: Other: Sham Acute intermittent hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia (AIH) — This will consist of up to 90 seconds of 9-10% O2 (FiO2 0.09), alternating with up to 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for a total of up to 45 minutes.
  Arms: AIH+ Upper extremity training; Acute intermittent hypoxia (AIH)
Behavioral: Upper extremity training — Subjects will receive 45 minutes of task-specific, high repetition upper extremity training, given using an upper-limb robotic rehabilitation device, the Armeo Spring®. Armeo Spring is a gravity support system based on an ergonomic arm exoskeleton with integrated springs. It cradles the entire arm, from shoulder to the hand, and counterbalances the weight of the user's arm. Therefore, it enhances any residual function and neuromuscular control, and assists in active movement across a large 3-D workspace. The Armeo software contains an extensive library of game-like movement exercises supported by a virtual-reality training environment that displays the functional task along with immediate performance feedback.
  Arms: AIH+ Upper extremity training; Sham AIH + Upper extremity training
Other: Sham Acute intermittent hypoxia — This will consist of up to 90 seconds of 21% O2 (FiO2 0.21), alternating with up to 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of alternating normoxic air will be repeated up to 18 times per session each, for a total of up to 45 minutes.
  Arms: Sham AIH + Upper extremity training; Sham Acute intermittent hypoxia

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a combinatorial therapy of breathing low oxygen in short bursts-acute intermittent hypoxia (AIH) and upper limb training on arm strength and function, and comparing it with individual treatments in persons with spinal cord injuries.

The investigators hypothesize that a combinatorial intervention with AIH therapy + upper limb training will be significantly more effective in improving hand function, compared to individual treatments alone.

To test this hypothesis, the investigators will determine the impact of combined daily AIH therapy and high-repetition task-specific upper extremity training on arm strength and hand dexterity in persons with spinal cord injuries.

DETAILED DESCRIPTION:
The objective of this research project is to determine the effect of a 5-day intervention with daily acute intermittent hypoxia (AIH) therapy, either alone or coupled with task-specific training, on upper extremity function in individuals with chronic, incomplete SCI.

Previous work already determined that breathing low levels of oxygen for short periods of time (also known as acute intermittent hypoxia) can improve lower limb motor function in persons with spinal injury. Specifically, this study is being done to determine if pre-treatment with intermittent hypoxia can enhance the beneficial effects of upper limb training on the restoration of limb function in persons with spinal injury.

This is a blinded study, which means that the subject will not know which treatment they are receiving. They will either receive intermittent periods of low oxygen (hypoxia) or a session composed of only normal room air. They will be randomly assigned to a treatment based on chance. Neither the subject nor the researcher chooses the assigned group. They will have an equal chance of being in either group.

The participant will receive a daily 5-day intervention with either acute intermittent hypoxia (AIH) therapy or room air, either alone or coupled with task-specific training, on upper extremity function in individuals with chronic, incomplete SCI. This will be preceded by a baseline testing visit prior to the intervention, and followed by a 4 week follow up period to assess the effects of the interventions over time.

The total duration of participation in the study intervention protocol is 1 week. Including the follow up period, the subjects will participate for a total of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Motor incomplete SCI at or below C2 and above T2 with non-progressive etiology
2. Age between 18 to 70 years
3. More than 1 year since SCI
4. Ability to close and open one's hand without assistance.
5. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Presence of any of the following medical conditions: congestive heart failure, arrhythmia, uncontrolled high blood pressure, uncontrolled diabetes mellitus, COPD/emphysema and severe asthma.
2. Weight over 250 pounds.
3. Persons with known coronary artery disease, a history of myocardial infarction and known carotid or intracerebral artery stenosis.
4. A medical clearance will be required if patients are taking any other investigational agents.
5. Women who are pregnant or nursing will be excluded, as the potential effects of intermittent hypoxia on pregnant women and fetus are unknown.
6. Individuals with tracheostomy will be excluded.
7. Subjects cannot pursue other research studies which may interfere with our treatment.
8. Subjects with diagnosed obstructive sleep apnea will be excluded as that may affect the response or sensitivity to AIH,
9. Orthopedic injuries or recent surgeries affecting the mobility of upper extremity and shoulder

We will not include the following populations:

* Adults unable to consent, unless accompanied by a legally authorized representative.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-24 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Grip strength (Hydraulic Handheld Dynamometer) | 10-12 minutes
  A dynamometer measures maximum gross grasp (kg) averaged over attempt with each hand. The minimum possible value of zero kg will be assigned when the participant cannot actively flex the fingers or grasp the dynamometer

SECONDARY OUTCOMES:
Pinch grip (Strength gauge Dynamometry) | 10-12 minutes
  A pinch gauge measures maximum pinch force (kg) averaged over attempt with each hand. The minimum possible value of zero kg will be assigned when the participant cannot actively squeeze the pinch meter between thumb and index finger.
Box and Block Test (BBT) | 5 min, with time to instruct
  Measure of manual dexterity that requires repeatedly moving 1-inch blocks from one side of a box to another in 60 seconds.
Nine Hole Peg Test | Upto 10-12 minutes, dependent on their ability to complete the test.
  A test of upper extremity dexterity which involves picking up pegs from a container and placing them, one by one, into holes on a board, as quickly as possible. Participants must then remove the pegs, one by one, and replace them into the original container. The total time in seconds is recorded.
Spinal Cord Independence Measure (SCIM III) | 10-15 minutes
  An outcome measure that is specifically designed to evaluate functional ability in individuals with spinal cord injury. It has established reliability, internal consistency, and construct validity (when compared to the Functional Independence Measure, and the Walking Index for Spinal Cord Injury). It consists of 19 items in 3 separate domains, including self-care, respiration and sphincter management, and mobility.
Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) | 45-60 minutes
  This is a clinical impairment measure used to evaluate sensory and motor hand function in individuals with cervical spinal cord injuries. It is composed of different domains, including: strength, sensation (dorsal and palmar), prehension ability, and prehension performance.
Capabilities of Upper Extremity Questionnaire | 10 minutes
  This is a structured interview that serves to evaluate functional limitations in individuals with tetraplegia. Participants are provided with questions regarding the difficulty of a given task as it relates to using their more-affected and less-affected sides. This outcome measure has established minimal detectable change and standard error of measure values. It also has demonstrated excellent criterion validity.
California Verbal Learning Test | 45 minutes
  The California Verbal Learning Test (CVLT) is a neuropsychological test which can be used to assess an individual's verbal memory abilities.
Delis-Kaplan Executive Function System (D-KEFS™) | 10-12 minutes
  Neurophysological test that assesses key components of executive functions within verbal and spatial modalities.
N-back test | 45 minutes
  The n -back task is a continuous performance task that is commonly used as an assessment in cognitive neuroscience to measure a part of working memory and working memory capacity.

CONTACTS AND LOCATIONS:
Overall Officials: William Z Rymer, MD, PhD, Study Director — Shirley Ryan AbilityLab; Milap Sandhu, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No